CLINICAL TRIAL: NCT04856670
Title: Assessing the Impact of Diabetes Mellitus on Anterior Chamber Cytokine Production and Postoperative Macular Edema in Patients Undergoing Femtosecond Laser-assisted Cataract Surgery
Brief Title: Assessing Diabetes Mellitus on Cytokine Analysis and Macular Edema Following FLACS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Uptown Eye Specialists (Other)
Responsible Party: Sponsor
Other Study IDs: UptownEye1
Record Dates: First submitted 2020-11-11; First posted 2021-04-23 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Cystoid Macular Edema; Diabetes Mellitus; Cataract
MeSH Terms: conditions — Macular Edema; Diabetes Mellitus; Cataract | interventions — Cataract Extraction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Control patients undergoing manual cataract surgery: As above
  Interventions: Procedure: Cataract surgery
- Control patients undergoing FLACS: Femtosecond laser assisted cataract surgery
  Interventions: Procedure: Cataract surgery
- Diabetic patients undergoing manual cataract surgery: As Above
  Interventions: Procedure: Cataract surgery
- diabetic patients undergoing FLACS: As Above
  Interventions: Procedure: Cataract surgery

INTERVENTIONS:
Procedure: Cataract surgery — Cataract surgery- Manual or femtosecond laser assisted

SUMMARY:
The purpose of this study is to assess the effects of diabetes mellitus (DM) on anterior chamber cytokine production and postoperative macular edema in patients undergoing femtosecond laser-assisted cataract surgery (FLACS). Patients with DM routinely undergo FLACS, yet the majority of studies evaluating intraocular inflammation following femtosecond laser treatment have excluded this patient population. Importantly, DM alters the inflammatory status of the eye, which may influence the production of inflammatory mediators following femtosecond laser treatment and the development of postoperative macular edema. The results from this study will provide insight into the risks and benefits of FLACS in patients with DM.

DETAILED DESCRIPTION:
As discussed above.

ELIGIBILITY:
Inclusion Criteria:

* All patients who are scheduled for manual cataract surgery or FLACS who have provided informed consent, in accordance with application regulations and guidelines.
* Only one eye from each participant will be included in the study (the first one to be operated on).

Exclusion Criteria:

* Intravitreal anti-VEGF injection < 3 months prior to cataract surgery
* Laser photocoagulation < 3 months prior to cataract surgery
* Complications during manual cataract surgery or FLACS
* Current or previous ocular or systemic inflammation
* History of rheumatic or immune disease
* Poor pharmacologic mydriasis
* Corneal opacities
* Pseudoexfoliation syndrome
* Previous ocular surgery or trauma
* Use of topical or systemic steroids < 6 months prior to surgery
* Prostaglandin analog eyedrop therapy
* Glaucoma
* Age-related macular degeneration

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients enrolling for Cataract surgery at Uptown Eye Specialists
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2021-05-25 (Estimated); Primary Completion 2021-09-15 (Estimated); Study Completion 2021-09-15 (Estimated)

PRIMARY OUTCOMES:
Aqueous humor concentrations of inflammatory mediators at the onset of manual cataract surgery and following femtosecond laser treatment | 1 day
  Cytokine concentration at time of cataract surgery

SECONDARY OUTCOMES:
Prevalence of postoperative macular edema in control and diabetic participants | Post op day 1, week 1, month 1 and month 3
  Macular edema post operatively
Postoperative change in central retinal thickness | Post op day 1, week 1, month 1 and month 3
  Central retinal thickness postoperatively
Postoperative change in macular volume | Post op day 1, week 1, month 1 and month 3
  macular volume postoperatively
Microvascular changes and development of cystic macular lesions | Post op day 1, week 1, month 1 and month 3
  Slit lamp exam of microvascular changes and development of cystic macular lesions
Best corrected visual acuity | Post op day 1, week 1, month 1 and month 3
  Change in visual acuity overtime
Prevalence and severity of postoperative flare | Post op day 1, week 1, month 1 and month 3
  Slit lamp exam for prevalence and severity of postoperative flare

CONTACTS AND LOCATIONS:
Overall Officials: sydney@emdi.ca Somani, MD, FRCSC, Principal Investigator — Uptown Eye Specialists
Locations (1):
- Uptown Eye Speicialists, Brampton, Otario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wu H, Hwang DK, Song X, Tao Y. Association between Aqueous Cytokines and Diabetic Retinopathy Stage. J Ophthalmol. 2017;2017:9402198. doi: 10.1155/2017/9402198. Epub 2017 Jun 7. PMID 28680705
- [Background] Dong N, Xu B, Wang B, Chu L, Tang X. Aqueous cytokines as predictors of macular edema in patients with diabetes following uncomplicated phacoemulsification cataract surgery. Biomed Res Int. 2015;2015:126984. doi: 10.1155/2015/126984. Epub 2015 Feb 25. PMID 25811020
- [Background] Agarwal A, Jacob S. Current and effective advantages of femto phacoemulsification. Curr Opin Ophthalmol. 2017 Jan;28(1):49-57. doi: 10.1097/ICU.0000000000000333. PMID 27801688
- [Background] Favuzza E, Becatti M, Gori AM, Mencucci R. Cytokines, chemokines, and flare in the anterior chamber after femtosecond laser-assisted cataract surgery. J Cataract Refract Surg. 2019 Jul;45(7):910-914. doi: 10.1016/j.jcrs.2019.01.040. PMID 31262481
- [Background] Liu YC, Setiawan M, Ang M, Yam GHF, Mehta JS. Changes in aqueous oxidative stress, prostaglandins, and cytokines: Comparisons of low-energy femtosecond laser-assisted cataract surgery versus conventional phacoemulsification. J Cataract Refract Surg. 2019 Feb;45(2):196-203. doi: 10.1016/j.jcrs.2018.09.022. Epub 2018 Dec 6. PMID 30528516
- [Background] Wang L, Zhang Z, Koch DD, Jia Y, Cao W, Zhang S. Anterior chamber interleukin 1beta, interleukin 6 and prostaglandin E2 in patients undergoing femtosecond laser-assisted cataract surgery. Br J Ophthalmol. 2016 Apr;100(4):579-82. doi: 10.1136/bjophthalmol-2015-307586. Epub 2015 Dec 11. PMID 26659713
- [Background] Chen H, Lin H, Zheng D, Liu Y, Chen W, Liu Y. Expression of Cytokines, Chmokines and Growth Factors in Patients Undergoing Cataract Surgery with Femtosecond Laser Pretreatment. PLoS One. 2015 Sep 2;10(9):e0137227. doi: 10.1371/journal.pone.0137227. eCollection 2015. PMID 26331724
- [Background] Chen H, Zhang X, Liao N, Wen F. Assessment of biomarkers using multiplex assays in aqueous humor of patients with diabetic retinopathy. BMC Ophthalmol. 2017 Oct 2;17(1):176. doi: 10.1186/s12886-017-0572-6. PMID 28969616
- [Background] Chu CJ, Johnston RL, Buscombe C, Sallam AB, Mohamed Q, Yang YC; United Kingdom Pseudophakic Macular Edema Study Group. Risk Factors and Incidence of Macular Edema after Cataract Surgery: A Database Study of 81984 Eyes. Ophthalmology. 2016 Feb;123(2):316-323. doi: 10.1016/j.ophtha.2015.10.001. Epub 2015 Dec 8. PMID 26681390
- [Derived] Cioana M, Patodia Y, Tong L, Chiu HH, Tam ES, Somani S. Anterior chamber cytokine production and postoperative macular edema in patients with diabetes undergoing FLACS. J Cataract Refract Surg. 2024 Feb 1;50(2):160-166. doi: 10.1097/j.jcrs.0000000000001335. PMID 37847109